CLINICAL TRIAL: NCT04044690
Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of IgPro20 (Subcutaneous Immunoglobulin, Hizentra®) in Adults With Dermatomyositis (DM) - The RECLAIIM Study
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of IgPro20 in Adults With Dermatomyositis (DM)
Acronym: RECLAIIM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Primary endpoint not attained
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IgPro20_3007; 2018-003171-35 (EudraCT Number); 2023-508293-28-00 (Other: EU CT Number)
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis | interventions — gamma-Globulins; Hizentra

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IgPro20 (Experimental): human immunoglobulin G administered subcutaneously
  Interventions: Drug: human immunoglobulin G
- Placebo (Placebo Comparator): human albumin solution administered subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: human immunoglobulin G — human immunoglobulin G administered subcutaneously
  Other Names: IgPro20; Hizentra
  Arms: IgPro20
Drug: Placebo — contains 2% human albumin, similar excipients as IgPro20 (Hizentra), same volume, same duration, administered subcutaneously
  Arms: Placebo

SUMMARY:
This is a phase 3, multicenter, randomized, placebo-controlled, double-blind study of IgPro20 (subcutaneous Ig) treatment in adult subjects with dermatomyositis (DM). The primary objective of this study is to assess the efficacy of IgPro20 subcutaneous (SC) doses in comparison to placebo in adult subjects with DM, as measured by responder status based on Total Improvement Score (TIS) assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age
* Diagnosis of at least probable idiopathic inflammatory myopathies (IIM) per European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) Classification Criteria which includes confirmation of dermatomyositis (DM) rash/manifestation, disease activity defined by presence of DM rash / manifestation or an objective disease activity measure
* Disease severity defined by Physician global activity visual analog scale (VAS) with a minimum value of 2.0 cm on a 10 cm scale and MMT-8 ≤ 142 or CDASI total activity score ≥ 14.
* Corticosteroid daily dose less than that or equal to 20 mg prednisolone equivalent

Exclusion Criteria:

* Cancer-associated myositis
* Evidence of active malignant disease or malignancies diagnosed within the previous 5 years
* Physician Global Damage score ≥ 3, or clinically relevant improvement between Screening Visit and Baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (76):
- United States (15):
  - 8401117 - Arizona Arthritis & Rheumatology Research, Glendale, Arizona
  - 8401199 - Neuromuscular Research Center, Phoenix, Arizona
  - 8401129 - UCLA - Rheumatology Los Angeles, Los Angeles, California
  - 8401473 - RecioMed Clinical Research Network, Inc., Boynton Beach, Florida
  - 8401160 - Center For Rheumatology, Fort Lauderdale, Florida
  - 8401132 - Omega Research Maitland, Orlando, Florida
  - 8401107 - Morsani Center for Advanced Health Care (CAHC), Tampa, Florida
  - 8401152 - The University of Kansas Medical Center, Fairway, Kansas
  - 8401476 - DS Research, Louisville, Kentucky
  - 8401487 - Ohio State University, Columbus, Ohio
  - 8401486 - Oregon Health and Science University, Portland, Oregon
  - 8401210 - University of Pennsylvania, Philadelphia, Pennsylvania
  - 8401151 - Biomedical Science Tower, Pittsburgh, Pennsylvania
  - 8401474 - West Tennessee Research Institute, LLC, Jackson, Tennessee
  - 8401115 - The University of Texas Medical School at Houston, Houston, Texas
- Argentina (4):
  - 0320083 - Hospital Italiano de Buenos Aires, Ciudad Autónoma Buenos Aires, Buenos Aires
  - 0320084 - DIM Clinica Privada, Buenos Aires
  - 0320081 - Fundacion Respirar, Buenos Aires
  - 0320077 - Centro Medico Privado de Reumatolgia, San Miguel de Tucumán
- Belgium (4):
  - 0560050 - Ghent Universit Hospital (UZ Gent), Ghent
  - 0560048 - Universitair Ziekenhuis (UZ) Leuven, Leuven
  - 0560056 - Universitair Ziekenhuis Leuven, Leuven
  - 0560049 - CHU de Liège - Sart Tilman, Liège
- France (6):
  - 2500146 - CHU De Dijon Hopital Du Bocage, Dijon
  - 2500188 - Centre Hospitalier Regional Universitaire de Lille, Lille
  - 2500133 - CHU - Hospital de la Timone, Marseille
  - 2500135 - CHU Nice-Hopital Archet I, Nice
  - 2500132 - Hopital Pitie-Salpetriere, Paris
  - 2500144 - Hopitaux Universitaire de Strasbourg, Strasbourg
- Germany (10):
  - 2760203 - Charité, Berlin
  - 2760211 - Charité - Universitätsmedizin Berlin, Berlin
  - 2760199 - University Hospital Köln, Cologne
  - 2760271 - Universitatsklinikum Carl Gustav Carus TU Dresden, Dresden
  - 2760273 - Hautklinik des Uni-Klinikums Erlangen, Erlangen
  - 2760036 - University Medicine Göttingen, Göttingen
  - 2760201 - Medizinische Hochschule Hannover (MHH), Hanover
  - 2760210 - University of Münster, Münster
  - 2760212 - University Hospital Of Tuebingen, Tübingen
  - 2760268 - University of Ulm, Ulm
- 3480048 - University of Debrecen, Debrecen, Hungary
- Italy (4):
  - 3800133 - Universita degli Studi Di Brescia - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - 3800132 - Universitaria Vittorio Emanuele, Catania
  - 3800139 - Universita degli Studi Firenze, Florence
  - 3800134 - Azienda Ospedaliero Universitaria Pisana, Pisa
- Japan (10):
  - 3920096 - Chukyo Hospital, Nagoya, Aichi-ken
  - 3920090 - University Of Fukui Hospital, Yoshida-Gun, Fukui
  - 3920088 - Gunma University Hospital, Maebashi, Gunma
  - 3920089 - Hokkaido University Hospital, Sapporo, Hokkaido
  - 3920086 - St. Marianna University Hospital, Kawasaki, Kanagawa
  - 3920125 - Tokyo Medical And Dental University Medical Hospital, Bunkyo, Tokyo
  - 3920091 - Nippon Medical School Hospital, Bunkyō-Ku, Tokyo
  - 3920097 - Tokyo Women's Medical University Hospital, Shinjuku-Ku, Tokyo
  - 3920087 - Wakayama Medical University Hospital, Wakayama
  - 3920035 - Yamaguchi University Hospital, Yamaguchi
- Mexico (3):
  - 4840081 - Centro Integral en Reumatologia, SA de CV, Guadalajara, Jalisco
  - 4840082 - CINTRE, Centro de Investigacion y Tratamiento Reumatologico S.C., Mexico City, Mexico City
  - 4840084 - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosí, S.C., San Luis Potosí City
- Poland (2):
  - 6160104 - Zespol Poradni Specjalistycznych REUMED, ONYKSOWA Filia nr 2, Lublin
  - 6160117 - MedicalConcierge Centrum Medyczne, Warsaw
- Russia (5):
  - 6430124 - ORIS Firm Limited Liability Company, Moscow
  - 6430122 - City Clinical Hospital No. 5, Nizhny Novgorod
  - 6430125 - Medical Centre-Healthy Family, Novosibirsk
  - 6430120 - St. Petersburg City Rheumatological Hospital 25, Saint Petersburg
  - 6430123 - Yaroslavl Oblast Clinical Hospital, Yaroslavl
- Spain (3):
  - 7240086 - Complejo Hospitalario Universitario A Coruña, A Coruña
  - 7240011 - Hospital Universitario Valle de Hebron, Barcelona
  - 7240112 - Hospital Clinic Barcelona, Barcelona
- Switzerland (2):
  - 7560033 - University Hospital Bern Inselspital, Bern
  - 7560028 - Kantonsspital St. Gallen, Sankt Gallen
- Ukraine (7):
  - 8040053 - Cherkassy Regional Hospital, Cherkasy
  - 8040055 - Mechnikov Institute of Microbiology and Immunology, Kharkiv
  - 8040057 - Khmelnitskiy Regional Hospital, Khmelnytskyi
  - 8040058 - State Institution National Scientific Center Strazhesko, Kiev
  - 8040052 - Institute of Rheumatology, Kyiv
  - 8040051 - Kyiv Railway Clinical Hospital No.2, Kyiv
  - 8040054 - Modern Clinic LLC, Zaporizhia

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 21 October 2019 to 02 December 2024.
Pre-assignment Details: A total of 199 participants were screened, and 65 of these were screen failures. A total of 134 were randomized in the study. This study consisted of 3 study periods (SP): SP1 (from Baseline to Week 25), SP2 (from Week 25 to 56) and SP3 (from Week 56 to approximately 5 years, study drug reimbursement was planned until drug becomes commercially available or if there is no longer benefit from the study drug). However, the study was terminated early.
Groups:
- Sequence A: IgPro20 / IgPro20 / IgPro20: Participants received IgPro20 subcutaneous (SC) infusions weekly for 24 weeks in Period 1, followed by IgPro20 SC infusions weekly for 28 weeks in Period 2. At Week 53, participants with demonstrated treatment benefit at Week 49 (Total Improvement Score [TIS] greater than or equal to (>=) 20 points) continued to Period 3 long-term treatment with open-label IgPro20 SC infusions weekly until the end of the study (EOS) (up to 5 years).
- Sequence B: Placebo / IgPro20 / IgPro20: Participants received matching placebo SC infusions weekly for 24 weeks in Period 1, followed by IgPro20 SC infusions weekly for 28 weeks in Period 2. At Week 53, participants with demonstrated treatment benefit at Week 49 (TIS >= 20 points) continued to Period 3 long-term treatment with open-label IgPro20 SC infusions weekly until the EOS (up to 5 years).
Period: Period 1
Arm/Group | Sequence A: IgPro20 / IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20 / IgPro20
Started | 67 | 67
Treated | 67 | 67
Completed | 56 | 55
Not Completed | 11 | 12
Not completed — Lack of Efficacy | 1 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Protocol Deviation | 2 | 0
Not completed — Site Terminated by Sponsor | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 1
Not completed — Death | 1 | 1
Not completed — Other: Unspecified | 1 | 0
Period: Period 2
Arm/Group | Sequence A: IgPro20 / IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20 / IgPro20
Started | 56 | 55
Treated | 56 | 55
Completed | 40 | 38
Not Completed | 16 | 17
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Site Terminated by Sponsor | 1 | 3
Not completed — Study Terminated by Sponsor | 8 | 3
Not completed — Death | 1 | 0
Not completed — Other: Unspecified | 1 | 1
Period: Period 3
Arm/Group | Sequence A: IgPro20 / IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20 / IgPro20
Started (Participants who completed SP2 and were eligible (TIS was >= 20 points at Week 49 visit) continued to SP3.) | 36 | 34
Treated | 36 | 34
Completed | 11 | 12
Not Completed | 25 | 22
Not completed — Site Terminated by Sponsor | 1 | 2
Not completed — Study Terminated by Sponsor | 24 | 18
Not completed — Missing | 0 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the safety (SAF) analysis set. The SAF analysis set comprised all participants who were randomized and received any amount of randomized investigational medicinal product (IMP) and were based on the actual treatment sequence received. Here, baseline characteristics are reported for Period 1, as participants from this cohort were selected to proceed to Periods 2 and 3.
Groups:
- IgPro20: Participants received IgPro20 SC infusions weekly for 24 weeks in Period 1.
- Placebo: Participants received matching placebo SC infusions weekly for 24 weeks in Period 1.
- Total: Total of all reporting groups
Arm/Group | IgPro20 | Placebo | Total
Number analyzed (Participants) | 67 | 67 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (15.86) | 49.1 (14.02) | 50.3 (14.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 51 | 98
  Male | 20 | 16 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 15 | 29
  Not Hispanic or Latino | 51 | 49 | 100
  Unknown or Not Reported | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 10 | 10 | 20
  Race: Black or African American | 3 | 1 | 4
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: White | 48 | 50 | 98
  Race: Other | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate
Description: A responder was defined as a participant with a TIS >= 20 points at Week 25 and at least 1 of the previous scheduled visits (Week 17 or 21), who completes 24 weeks of randomized IMP treatment without the use of rescue corticosteroid treatment. The TIS was a sum response criterion which incorporates 6 weighted international myositis assessment and clinical studies (IMACS) core set measures (CSMs) including Physician and Patient Global Disease Activity (PGA), Manual Muscle Testing-8 (MMT-8), Health Assessment Questionnaire, Muscle Enzyme, and Extramuscular Global Activity (EGA). Thresholds for minimal, moderate, and major improvement were >= 20, >= 40, and >= 60 points, respectively on the TIS. Percentage of responders at Week 25 based on TIS are reported here. Multiple imputation (MI) was used to impute missing values for participants who discontinued due to the military activities in Ukraine.
Time Frame: At Week 25
Population: Analysis was performed on the modified intent-to-treat (mITT) analysis set. The mITT analysis set comprises all participants who underwent study screening procedures, were randomized to receive any amount of randomized IMP. The documented failure to take any amount of randomized IMP or the lack of any post randomization efficacy data lead to the exclusion of the participant from the mITT.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
percentage of participants | 64.3 [52.56 to 75.99] | 61.6 [49.52 to 73.74]
Statistical Analysis 1: Comparison: IgPro20 vs Placebo; Test type: Superiority; p = 0.371008, Regression, Logistic — Threshold of significance at <= 0.025; Exact logistic regression model including fixed effects for treatment, region (Japan vs. non-Japan) and Baseline MMT-8 (≤ 142 points vs. >142 points); Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.551 to 2.309] — Rubin's rule applied following MI

2. Secondary Outcome: Mean TIS
Description: The TIS was a sum response criterion which incorporates 6 weighted IMACS CSMs including Physician and PGA, MMT-8, Health Assessment Questionnaire, Muscle Enzyme, and EGA. A total improvement score (range 0 to 100; higher the score, better the condition), determined by summing scores for each CSM, was based on improvement in and relative weight of each CSM. Thresholds for minimal, moderate, and major improvement were >= 20, >= 40, and >= 60 points, respectively on the TIS. Least squares (LS) means were estimated using a mixed model repeated measures (MMRM) including treatment, visit, the interaction between treatment and visit, region, and baseline MMT-8 (<=142 points vs >142 points) as fixed effects, participant as a random effect.
Time Frame: At Week 25
Population: Analysis was performed on the mITT analysis set. The mITT analysis set comprises all participants who underwent study screening procedures and were randomized to receive any amount of randomized IMP. The documented failure to take any amount of randomized IMP, or the lack of any post-randomization efficacy data, led to the exclusion of the participant from the mITT.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
score on a scale | 32.24 [25.275 to 39.208] | 30.78 [23.668 to 37.896]
Statistical Analysis 1: Comparison: IgPro20 vs Placebo; Test type: Superiority; p = 0.360939, MMRM — Descriptive p-value; LS mean difference = 1.46, 95% CI 2-sided [-6.651 to 9.570]

3. Secondary Outcome: Mean Changes From Baseline in MMT-8
Description: The MMT-8 was a set of 8 designated muscles which were tested bilaterally (potential score ranging from 0 to 150): 7 biaxial muscles with a potential score 0 to 140 and 1 axial (neck flexors) with a potential score of 0 to 10. Improvement is documented with an increase in score. LS means were estimated using a MMRM including treatment, visit, the interaction between treatment and visit, and region as fixed effects, baseline MMT-8 as a continuous covariate and participant as a random effect.
Time Frame: From Baseline to Week 25
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
score on a scale | 8.9 [4.08 to 13.78] | 11.3 [4.79 to 17.89]
Statistical Analysis 1: Comparison: IgPro20 vs Placebo; Test type: Superiority; p = 0.730994, MMRM — Descriptive p-value; LS mean difference = -2.4, 95% CI 2-sided [-10.15 to 5.33]

4. Secondary Outcome: Mean Changes From Baseline in Cutaneous Dermatomyositis Disease Area and Severity Index Total Activity Score (CDASI-A)
Description: The CDASI in its modified version 2 (V2) is a validated tool of skin disease activity (3 items) and damage (3 items) assessment. Scores range from 0-100 for activity and from 0-32 for damage. Improvement is documented with a decrease in score. LS means were estimated using a MMRM including treatment, visit, the interaction between treatment and visit, region, and baseline MMT-8 (<=142 points vs >142 points) as fixed effects, baseline CDASI-A as a continuous covariate, and participants as a random effect.
Time Frame: From Baseline to Week 25
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
score on a scale | -10.6 [-13.28 to -7.82] | -5.3 [-8.29 to -2.28]
Statistical Analysis 1: Comparison: IgPro20 vs Placebo; Test type: Superiority; p = 0.001647, MMRM — Descriptive p-value; LS mean difference = -5.3, 95% CI 2-sided [-8.72 to -1.82]

5. Secondary Outcome: Percentage of Participants Who Are Able to Reduce the Oral Corticosteroid Dose by >= 25%
Description: Reduction in corticosteroid dose.
Time Frame: At Week 25
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
percentage of participants | 23.2 [12.89 to 33.45] | 20.2 [10.39 to 30.04]
Statistical Analysis 1: Comparison: IgPro20 vs Placebo; Test type: Superiority; p = 0.335347, Regression, Logistic — Descriptive p-value; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.520 to 2.766] — Rubin's rule for combination applied following MI

6. Secondary Outcome: Period 1: Mean TIS at Each Visit
Description: The TIS was a sum response criterion which incorporates 6 weighted IMACS CSMs including Physician and PGA, MMT-8, Health Assessment Questionnaire, Muscle Enzyme, and EGA. A total improvement score (range 0 to 100), determined by summing scores for each CSM, was based on improvement in and relative weight of each CSM. Thresholds for minimal, moderate, and major improvement were >= 20, >= 40, and >= 60 points on the TIS.
Time Frame: At Week 5, 9, 13, 17, 21, and 25
Population: Analysis was performed on the mITT analysis set. Here, overall number of participants analyzed (N) = participants evaluable for this outcome measure, and number analyzed (n) = participants with evaluable data for each specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 59 | 62
score on a scale
  Week 5 | 23.22 (16.387) | 20.97 (16.684)
  Week 9: number analyzed (Participants) | 59 | 57
  Week 9 | 32.54 (18.132) | 26.67 (17.924)
  Week 13: number analyzed (Participants) | 56 | 55
  Week 13 | 37.68 (17.267) | 31.68 (20.705)
  Week 17: number analyzed (Participants) | 55 | 51
  Week 17 | 41.00 (16.926) | 35.44 (21.458)
  Week 21: number analyzed (Participants) | 54 | 48
  Week 21 | 43.56 (17.112) | 36.67 (21.882)
  Week 25: number analyzed (Participants) | 51 | 47
  Week 25 | 40.20 (20.093) | 40.21 (21.812)

7. Secondary Outcome: Period 2: Mean TIS at Each Visit
Description: as for outcome 6
Time Frame: Week 25, 29, 33, 37, 41, 45, 49, and 53
Population: Analysis was performed on the mITT analysis set extended (mITT-Ex) that comprised all participants in mITT who completed the first 24 weeks of SP1 and received any amount of the IMP in SP2. The documented failure to take any amount of randomized IMP in SP2 led to the exclusion of the participant from mITT-Ex. Here, overall number of participants analyzed (N) = participants evaluable for this outcome measure, and number analyzed (n) = participants with evaluable data for each specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sequence A: IgPro20 / IgPro20: Participants received IgPro20 SC infusions weekly for 24 weeks in Period 1, followed by IgPro20 SC infusions weekly for 28 weeks in Period 2.
- Sequence B: Placebo / IgPro20: Participants received matching placebo SC infusions weekly for 24 weeks in Period 1, followed by IgPro20 SC infusions weekly for 28 weeks in Period 2.
Arm/Group | Sequence A: IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20
Number analyzed (Participants) | 54 | 52
score on a scale
  Week 25 | 40.09 (19.547) | 38.08 (22.658)
  Week 29: number analyzed (Participants) | 53 | 52
  Week 29 | 45.05 (19.931) | 42.74 (20.057)
  Week 33: number analyzed (Participants) | 51 | 51
  Week 33 | 44.66 (19.346) | 46.23 (18.258)
  Week 37: number analyzed (Participants) | 48 | 48
  Week 37 | 47.81 (18.805) | 48.49 (17.071)
  Week 41: number analyzed (Participants) | 46 | 46
  Week 41 | 50.49 (18.255) | 51.68 (15.943)
  Week 45: number analyzed (Participants) | 45 | 45
  Week 45 | 50.89 (19.018) | 52.94 (15.078)
  Week 49: number analyzed (Participants) | 43 | 39
  Week 49 | 51.63 (17.844) | 50.51 (16.010)
  Week 53: number analyzed (Participants) | 39 | 37
  Week 53 | 50.32 (15.886) | 54.26 (15.022)

8. Secondary Outcome: Period 1: Percentage of Participants Achieving TIS ≥ 20, ≥ 40 and ≥ 60 Points
Description: Participants were considered and reported in more than one category (TIS >= 20, >= 40 and >= 60 Points).
Time Frame: At Week 5, 9, 13, 17, 21, and 25
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
percentage of participants
  Week 5: TIS >= 20 Points | 47.7 [35.15 to 60.46] | 47.7 [35.15 to 60.46]
  Week 5: TIS >= 40 Points | 16.9 [8.76 to 28.27] | 15.4 [7.63 to 26.48]
  Week 5: TIS >= 60 Points | 1.5 [0.04 to 8.28] | 1.5 [0.04 to 8.28]
  Week 9: TIS >= 20 Points | 63.1 [50.20 to 74.72] | 56.3 [43.28 to 68.63]
  Week 9: TIS >= 40 Points | 32.3 [21.23 to 45.05] | 26.6 [16.30 to 39.09]
  Week 9: TIS >= 60 Points | 9.2 [3.46 to 19.02] | 4.7 [0.98 to 13.09]
  Week 13: TIS >= 20 Points | 73.8 [61.46 to 83.97] | 60.9 [47.93 to 72.90]
  Week 13: TIS >= 40 Points | 36.9 [25.28 to 49.80] | 31.3 [20.24 to 44.06]
  Week 13: TIS >= 60 Points | 13.8 [6.53 to 24.66] | 10.9 [4.51 to 21.25]
  Week 17: TIS >= 20 Points | 75.4 [63.13 to 85.23] | 57.8 [44.82 to 70.06]
  Week 17: TIS >= 40 Points | 44.6 [32.27 to 57.47] | 34.4 [22.95 to 47.30]
  Week 17: TIS >= 60 Points | 15.4 [7.63 to 26.48] | 15.6 [7.76 to 26.86]
  Week 21: TIS >= 20 Points | 73.4 [60.91 to 83.70] | 60.3 [47.20 to 72.43]
  Week 21: TIS >= 40 Points | 53.1 [40.23 to 65.72] | 33.3 [21.95 to 46.34]
  Week 21: TIS >= 60 Points | 18.8 [10.08 to 30.46] | 12.7 [5.65 to 23.50]
  Week 25: TIS >= 20 Points | 64.1 [51.10 to 75.68] | 65.1 [52.03 to 76.66]
  Week 25: TIS >= 40 Points | 45.3 [32.82 to 58.25] | 39.7 [27.57 to 52.80]
  Week 25: TIS >= 60 Points | 17.2 [8.90 to 28.68] | 15.9 [7.88 to 27.26]

9. Secondary Outcome: Period 2: Percentage of Participants Achieving TIS ≥ 20, ≥ 40 and ≥ 60 Points
Description: Participants were considered and reported in more than one category (TIS >= 20, >= 40 and >= 60 Points).
Time Frame: Week 25, 29, 33, 37, 41, 45, 49, and 53
Population: Analysis was performed on the mITT-Ex analysis set. The mITT-Ex comprised all participants in mITT who completed the first 24 weeks of SP1 and received any amount of the IMP in SP2. The documented failure to take any amount of randomized IMP in SP2 led to the exclusion of the participant from mITT-Ex.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sequence A: IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20
Number analyzed (Participants) | 55 | 54
percentage of participants
  Week 25: TIS >= 20 Points | 80.0 [67.03 to 89.57] | 77.8 [64.40 to 87.96]
  Week 25: TIS >= 40 Points | 56.4 [42.32 to 69.70] | 48.1 [34.34 to 62.16]
  Week 25: TIS >= 60 Points | 20.0 [10.43 to 32.97] | 18.5 [9.25 to 31.43]
  Week 29: TIS >= 20 Points | 87.0 [75.10 to 94.63] | 84.9 [72.41 to 93.25]
  Week 29: TIS >= 40 Points | 64.8 [50.62 to 77.32] | 54.7 [40.45 to 68.44]
  Week 29: TIS >= 60 Points | 31.5 [19.52 to 45.55] | 22.6 [12.28 to 36.21]
  Week 33: TIS >= 20 Points | 85.2 [72.88 to 93.38] | 90.6 [79.34 to 96.87]
  Week 33: TIS >= 40 Points | 57.4 [43.21 to 70.77] | 64.2 [49.80 to 76.86]
  Week 33: TIS >= 60 Points | 22.2 [12.04 to 35.60] | 24.5 [13.76 to 38.28]
  Week 37: TIS >= 20 Points | 82.7 [69.67 to 91.77] | 88.5 [76.56 to 95.65]
  Week 37: TIS >= 40 Points | 57.7 [43.20 to 71.27] | 67.3 [52.89 to 79.67]
  Week 37: TIS >= 60 Points | 28.8 [17.13 to 43.08] | 25.0 [14.03 to 38.95]
  Week 41: TIS >= 20 Points | 84.3 [71.41 to 92.98] | 84.6 [71.92 to 93.12]
  Week 41: TIS >= 40 Points | 64.7 [50.07 to 77.57] | 73.1 [58.98 to 84.43]
  Week 41: TIS >= 60 Points | 37.3 [24.13 to 51.92] | 30.8 [18.72 to 45.10]
  Week 45: TIS >= 20 Points | 80.0 [66.28 to 89.97] | 84.3 [71.41 to 92.98]
  Week 45: TIS >= 40 Points | 64.0 [49.19 to 77.08] | 66.7 [52.08 to 79.24]
  Week 45: TIS >= 60 Points | 40.0 [26.41 to 54.82] | 31.4 [19.11 to 45.89]
  Week 49: TIS >= 20 Points | 80.0 [66.28 to 89.97] | 70.0 [55.39 to 82.14]
  Week 49: TIS >= 40 Points | 68.0 [53.30 to 80.48] | 58.0 [43.21 to 71.81]
  Week 49: TIS >= 60 Points | 36.0 [22.92 to 50.81] | 22.0 [11.53 to 35.96]
  Week 53: TIS >= 20 Points | 78.0 [64.04 to 88.47] | 72.0 [57.51 to 83.77]
  Week 53: TIS >= 40 Points | 56.0 [41.25 to 70.01] | 66.0 [51.23 to 78.79]
  Week 53: TIS >= 60 Points | 30.0 [17.86 to 44.61] | 24.0 [13.06 to 38.17]

10. Secondary Outcome: Period 1: Time to First Achieving TIS >= 20, >= 40, and >= 60 Points on the TIS
Description: The observation was censored if no improvement was observed before the intake of rescue/increased doses of oral corticosteroids in SP1 or before the end of the period.
Time Frame: Up to Week 25
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
days
  TIS >= 20 Points | 31.0 [28.00 to 56.00] | 32.0 [28.00 to 56.00]
  TIS >= 40 Points | 112.0 [63.00 to 141.00] | 112.0 [84.00 to 168.00]
  TIS >= 60 Points | NA [NA to NA] — Median and 95% CI are not estimable due to an insufficient number of participants with event (TIS >= 60 points), due to a high number of censored observations. | NA [170.00 to NA] — Median and upper limit of 95% CI are not estimable due to an insufficient number of participants with event (TIS >= 60 points), due to a high number of censored observations.

11. Secondary Outcome: Period 1 and 2: Time to First Achieving TIS >= 20, >= 40, and >= 60 Points Improvement on the TIS
Description: as for outcome 10
Time Frame: Up to Week 53
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sequence A: IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20
Number analyzed (Participants) | 65 | 65
days
  TIS >= 20 Points | 31.0 [28.00 to 56.00] | 32.0 [28.00 to 56.00]
  TIS >= 40 Points | 112.0 [63.00 to 141.00] | 137.0 [84.00 to 196.00]
  TIS >= 60 Points | 308.0 [196.00 to NA] — Upper limit of CI was not estimable due to an insufficient number of participants with event (TIS >= 60 points), due to a high number of censored observations. | 336.0 [249.00 to NA] — Upper limit of CI was not estimable due to an insufficient number of participants with event (TIS >= 60 points), due to a high number of censored observations.

12. Secondary Outcome: Mean Changes From Baseline in Individual CSMs (Except Muscle Enzymes) and CDASI
Description: Individual CSMs included following: Myositis Disease Activity Assessment Tool (MDAAT) Physician global disease activity (PGDA), PGA assessment, MMT-8, health assessment questionnaire-disability index (HAQ-DI), and MDAAT-EGA. Higher values were associated with a better state of health for the MMT-8 (range 0 -150) assessment, while lower values were associated with a better state of health for: MDAAT-PGDA (range 0 -100), PGA (range 0-100), HAQ-DI (range 0-3), MDAAT-EGA (range 0 -100), and CDASI-A (range 0-100).
Time Frame: From Baseline to Week 25
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 52 | 48
score on a scale
  MMT-8: Week 25: number analyzed (Participants) | 51 | 47
  MMT-8: Week 25 | 10.8 (16.71) | 15.2 (24.02)
  MDAAT-PGDA: Week 25: number analyzed (Participants) | 51 | 47
  MDAAT-PGDA: Week 25 | -21.2 (19.86) | -21.8 (18.64)
  MDAAT-EGA: Week 25: number analyzed (Participants) | 51 | 47
  MDAAT-EGA: Week 25 | -17.4 (22.54) | -13.9 (17.67)
  PGA: Week 25 | -13.0 (26.52) | -16.8 (20.57)
  HAQ - DI: Week 25 | -0.195 (0.4627) | -0.172 (0.4801)
  CDASI-A: Week 25: number analyzed (Participants) | 51 | 47
  CDASI-A: Week 25 | -11.5 (10.85) | -7.9 (8.91)

13. Secondary Outcome: Mean Changes From Week 25 in Individual CSMs (Except Muscle Enzymes) and CDASI
Description: Individual CSMs included following: MDAAT-PGDA, PGA assessment, MMT-8, HAQ-DI, and MDAAT extramacular global assessment. Higher values were associated with a better state of health for the MMT-8 (range 0 -150) assessment, while lower values were associated with a better state of health for: MDAAT-PGDA (range 0 -100), PGA (range 0-100), HAQ-DI (range 0-3), MDAAT-EGA (range 0 -100), and CDASI-A (range 0-100).
Time Frame: From Week 25 to Week 53
Population: Analysis was performed on the mITT-Ex analysis set. The mITT-Ex comprised all participants in mITT who completed the first 24 weeks of SP1 and received any amount of the IMP in SP2. The documented failure to take any amount of randomized IMP in SP2 led to the exclusion of the participant from mITT-Ex. Here, overall number of participants analyzed (N) = participants evaluable for this outcome measure, and number analyzed (n) = participants with evaluable data for each specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sequence A: IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20
Number analyzed (Participants) | 40 | 37
score on a scale
  MMT-8: Week 53: number analyzed (Participants) | 39 | 36
  MMT-8: Week 53 | 7.1 (11.32) | 7.9 (13.44)
  MDAAT-PGDA: Week 53: number analyzed (Participants) | 39 | 36
  MDAAT-PGDA: Week 53 | -8.5 (17.13) | -15.5 (18.74)
  MDAAT-EGA: Week 53: number analyzed (Participants) | 39 | 36
  MDAAT-EGA: Week 53 | -0.9 (12.38) | -11.5 (18.21)
  PGA: Week 53 | -3.3 (20.94) | -9.0 (23.87)
  HAQ - DI: Week 53 | -0.106 (0.2587) | -0.162 (0.4477)
  CDASI-A: Week 53: number analyzed (Participants) | 39 | 36
  CDASI-A: Week 53 | -0.8 (7.52) | -5.3 (9.70)

14. Secondary Outcome: Period 1: Number of Participants Meeting Definition of Worsening (DOW) at Least Once, Twice, or > Twice
Description: The DOW consists of meeting 1 of the following criteria on 2 consecutive visits at least 2 weeks apart: PGA Assessment Visual Analog Scale (VAS) worsening >= 2 cm* and MMT-8 worsening >= absolute 10%, or EGA worsening >= 2 cm on the MDAAT VAS, or Any 3 of 6 CSM worsening by >= absolute 20%. (*If baseline PGA VAS is 8 to 10, then any worsening on Physician Global VAS was acceptable as long as MMT-8 criterion was met.)
Time Frame: Up to Week 25
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
Participants
  At Least Once | 2 | 3
  At Least Twice | 0 | 0
  More Than Twice | 0 | 0

15. Secondary Outcome: Period 1: Percentage of Participants Meeting DOW at Least Once, Twice, or > Twice
Description: The DOW consists of meeting 1 of the following criteria on 2 consecutive visits at least 2 weeks apart: PGA Assessment VAS worsening >= 2 cm* and MMT-8 worsening >= absolute 10%, or EGA worsening >= 2 cm on the MDAAT VAS, or Any 3 of 6 CSM worsening by >= absolute 20%. (*If baseline PGA VAS is 8 to 10, then any worsening on Physician Global VAS was acceptable as long as MMT-8 criterion was met.)
Time Frame: Up to Week 25
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
percentage of participants
  At Least Once | 3.1 | 4.6
  At Least Twice | 0 | 0
  More Than Twice | 0 | 0

16. Secondary Outcome: Period 2: Number of Participants Meeting DOW at Least Once, Twice, or > Twice
Description: as for outcome 15
Time Frame: From Week 25 up to Week 53
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20
Number analyzed (Participants) | 55 | 54
Participants
  At Least Once | 2 | 1
  At Least Twice | 0 | 0
  More Than Twice | 0 | 0

17. Secondary Outcome: Period 2: Percentage of Participants Meeting DOW at Least Once, Twice, or > Twice
Description: as for outcome 15
Time Frame: From Week 25 up to Week 53
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A: IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20
Number analyzed (Participants) | 55 | 54
percentage of participants
  At Least Once | 3.6 | 1.9
  At Least Twice | 0 | 0
  More Than Twice | 0 | 0

18. Secondary Outcome: Time to Meeting DOW for the First Time
Description: The DOW consists of meeting 1 of the following criteria on 2 consecutive visits at least 2 weeks apart: PGA Assessment VAS worsening >= 2 cm* and MMT-8 worsening >= absolute 10%, or EGA worsening >= 2 cm on the MDAAT VAS, or Any 3 of 6 CSM worsening by >= absolute 20%. (*If baseline PGA VAS is 8 to 10, then any worsening on Physician Global VAS was acceptable as long as MMT-8 criterion was met.) The observation was censored if no DOW was observed before the intake of rescue treatment or before the end of the period.
Time Frame: Up to Week 53
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sequence A: IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20
Number analyzed (Participants) | 65 | 65
days | NA [NA to NA] — Median and 95% CI are not estimable due to an insufficient number of participants with event (DOW), due to a high number of censored observations. | NA [NA to NA] — Median and 95% CI are not estimable due to an insufficient number of participants with event (DOW), due to a high number of censored observations.

19. Secondary Outcome: Number of Participants Meeting DOW and Receiving Rescue Steroid Treatment
Description: The DOW consists of meeting 1 of the following criteria on 2 consecutive visits at least 2 weeks apart: PGA Assessment VAS worsening >= 2 cm* and MMT-8 worsening >= absolute 10%, or EGA worsening >= 2 cm on the MDAAT VAS, or Any 3 of 6 CSM worsening by >= absolute 20%. (*If baseline PGA VAS is 8 to 10, then any worsening on Physician Global VAS was acceptable as long as MMT-8 criterion was met.) The Number of participants meeting DOW and who received rescue steroid treatment are reported here.
Time Frame: Up to Week 25
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
Participants | 0 | 2

20. Secondary Outcome: Percentage of Participants Meeting DOW and Receiving Rescue Steroid Treatment
Description: The DOW consists of meeting 1 of the following criteria on 2 consecutive visits at least 2 weeks apart: PGA Assessment VAS worsening >= 2 cm* and MMT-8 worsening >= absolute 10%, or EGA worsening >= 2 cm on the MDAAT VAS, or Any 3 of 6 CSM worsening by >= absolute 20%. (*If baseline PGA VAS is 8 to 10, then any worsening on Physician Global VAS was acceptable as long as MMT-8 criterion was met.) The percentage of participants meeting DOW and who received rescue steroid treatment are reported here.
Time Frame: Up to Week 25
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
percentage of participants | 0 | 3.1

21. Secondary Outcome: Number of Participants Who Start Oral Corticosteroid Dose Taper
Time Frame: Up to Week 25
Population: Analysis was performed on the mITT analysis set. The mITT analysis set comprises all participants who underwent study screening procedures and were randomized to receive any amount of randomized IMP. The documented failure to take any amount of randomized IMP, or the lack of any post-randomization efficacy data, led to the exclusion of the participant from the mITT. Here, overall number of participants analyzed (N) = participants with oral concomitant corticosteroid treatment at Week 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 46 | 48
Participants | 19 | 19

22. Secondary Outcome: Percentage of Participants Who Start Oral Corticosteroid Dose Taper
Time Frame: Up to Week 25
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 46 | 48
percentage of participants | 41.3 | 39.6

23. Secondary Outcome: Number of Participants Who Are Able to Reduce the Oral Corticosteroid Dose by >= 25%, >= 50%, >= 75%
Time Frame: Up to Week 25 and 52
Population: Analysis was performed on the mITT-Ex analysis set. The mITT-Ex comprised all participants in mITT who completed the first 24 weeks of SP1 and received any amount of the IMP in SP2. The documented failure to take any amount of randomized IMP in SP2 led to the exclusion of the participant from mITT-Ex. Here, overall number of participants analyzed (N) = all participants with oral concomitant corticosteroid treatment at Week 1 who were part of mITT Ex.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20
Number analyzed (Participants) | 40 | 39
Participants
  Week 25: Reduction >= 25% | 16 | 14
  Week 25: Reduction >= 50% | 11 | 8
  Week 25: Reduction >= 75% | 3 | 3
  Week 52: Reduction >= 25% | 19 | 17
  Week 52: Reduction >= 50% | 17 | 14
  Week 52: Reduction >= 75% | 12 | 9

24. Secondary Outcome: Percentage of Participants Who Are Able to Reduce the Oral Corticosteroid Dose by >= 25%, >= 50%, >= 75%
Time Frame: Up to Week 25 and 52
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A: IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20
Number analyzed (Participants) | 40 | 39
percentage of participants
  Week 25: Reduction >= 25% | 40.0 | 35.9
  Week 25: Reduction >= 50% | 27.5 | 20.5
  Week 25: Reduction >= 75% | 7.5 | 7.7
  Week 52: Reduction >= 25% | 47.5 | 43.6
  Week 52: Reduction >= 50% | 42.5 | 35.9
  Week 52: Reduction >= 75% | 30.0 | 23.1

25. Secondary Outcome: Percentage of Participants Receiving Rescue Corticosteroid Treatment
Time Frame: Up to Week 25
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
percentage of participants | 1.5 | 9.2

26. Secondary Outcome: Percentage of Participants Whose Rescue Corticosteroid Treatment is Tapered
Time Frame: Up to Week 25
Population: Analysis was performed on the mITT analysis set. The mITT analysis set comprises all participants who underwent study screening procedures and were randomized to receive any amount of randomized IMP. The documented failure to take any amount of randomized IMP, or the lack of any post-randomization efficacy data, led to the exclusion of the participant from the mITT. Here, overall number of participants analyzed (N) = participants receiving oral rescue corticosteroid treatment up to Week 25.
Measure: Number; unit: percentage of participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 1 | 6
percentage of participants | 0 | 100.0

27. Secondary Outcome: Time to First Intake of Rescue Corticosteroid Treatment
Description: The observation was censored if no Rescue was observed before the last day of the last week with IMP intake or before the end of the period.
Time Frame: Up to Week 25
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 65 | 65
days | NA [NA to NA] — Median and 95% CI are not estimable due to an insufficient number of participants with event (intake of rescue treatment), due to a high number of censored observations. | NA [NA to NA] — Median and 95% CI are not estimable due to an insufficient number of participants with event (intake of rescue treatment), due to a high number of censored observations.

28. Secondary Outcome: Number of Participants Having at Least 1 Level, 2 Levels, and More Than 2 Levels of Improvement From Baseline in Mobility, Self-care, and Usual Activities Domains of EuroQoL 5-Dimension Questionnaire (EQ-5D-5L)
Description: EQ-5D-5L was assessed across 5 levels, with participants selecting the option that best described their health on that day, ranging from "no problems" to "unable to" walk, wash/dress, or perform usual activities. Out of total participants of each arm, only participants having at least 1 Level, 2 Levels, and more than 2 Levels of improvement from baseline in Mobility, Self-care, and Usual Activities Domains of EQ-5D-5L are reported in this outcome measure.
Time Frame: From Baseline to Week 13 and 25
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 57 | 55
Participants
  Week 13: Mobility: At least 1 level improvement | 16 | 15
  Week 13: Mobility: At least 2 level improvement | 1 | 0
  Week 13: Mobility: More than 2 level improvement | 0 | 0
  Week 13: Self-Care: At least 1 level improvement | 15 | 13
  Week 13: Self-Care: At least 2 level improvement | 2 | 2
  Week 13: Self-Care: More than 2 level improvement | 1 | 0
  Week 13: Usual Activities: At least 1 level improvement | 16 | 15
  Week 13: Usual Activities: At least 2 level improvement | 1 | 3
  Week 13: Usual Activities: More than 2 level improvement | 1 | 0
  Week 25: Mobility: At least 1 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Mobility: At least 1 level improvement | 10 | 14
  Week 25: Mobility: At least 2 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Mobility: At least 2 level improvement | 5 | 3
  Week 25: Mobility: More than 2 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Mobility: More than 2 level improvement | 0 | 0
  Week 25: Self-Care: At least 1 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Self-Care: At least 1 level improvement | 9 | 15
  Week 25: Self-Care: At least 2 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Self-Care: At least 2 level improvement | 2 | 3
  Week 25: Self-Care: More than 2 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Self-Care: More than 2 level improvement | 2 | 0
  Week 25: Usual Activities: At least 1 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Usual Activities: At least 1 level improvement | 15 | 13
  Week 25: Usual Activities: At least 2 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Usual Activities: At least 2 level improvement | 2 | 1
  Week 25: Usual Activities: More than 2 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Usual Activities: More than 2 level improvement | 1 | 0

29. Secondary Outcome: Percentage of Participants Having at Least 1 Level, 2 Levels, and More Than 2 Levels of Improvement From Baseline in Mobility, Self-care, and Usual Activities Domains of EQ-5D-5L
Description: as for outcome 28
Time Frame: From Baseline to Week 13 and 25
Population: Analysis was performed on the mITT analysis set. Here, overall number of participants analyzed (N) = participants evaluable for this outcome measure, and number analyzed (n) = participants with evaluable data for each specified category.
Measure: Number; unit: percentage of participants
Arm/Group | IgPro20 | Placebo
Number analyzed (Participants) | 57 | 55
percentage of participants
  Week 13: Mobility : At least 1 level improvement | 28.1 | 27.3
  Week 13: Mobility : At least 2 level improvement | 1.8 | 0
  Week 13: Mobility : More than 2 level improvement | 0 | 0
  Week 13: Self-Care : At least 1 level improvement | 26.3 | 23.6
  Week 13: Self-Care : At least 2 level improvement | 3.5 | 3.6
  Week 13: Self-Care : More than 2 level improvement | 1.8 | 0
  Week 13: Usual Activities : At least 1 level improvement | 28.1 | 27.3
  Week 13: Usual Activities : At least 2 level improvement | 1.8 | 5.5
  Week 13: Usual Activities : More than 2 level improvement | 1.8 | 0
  Week 25: Mobility : At least 1 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Mobility : At least 1 level improvement | 19.2 | 29.2
  Week 25: Mobility : At least 2 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Mobility : At least 2 level improvement | 9.6 | 6.3
  Week 25: Mobility : More than 2 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Mobility : More than 2 level improvement | 0 | 0
  Week 25: Self-Care : At least 1 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Self-Care : At least 1 level improvement | 3.8 | 31.3
  Week 25: Self-Care : At least 2 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Self-Care : At least 2 level improvement | 1.9 | 6.3
  Week 25: Self-Care : More than 2 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Self-Care : More than 2 level improvement | 1.9 | 0
  Week 25: Usual Activities : At least 1 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Usual Activities : At least 1 level improvement | 15.8 | 29.3
  Week 25: Usual Activities : At least 2 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Usual Activities : At least 2 level improvement | 5.3 | 5.2
  Week 25: Usual Activities : More than 2 level improvement: number analyzed (Participants) | 52 | 48
  Week 25: Usual Activities : More than 2 level improvement | 3.5 | 0

30. Secondary Outcome: Number of Participants Having no Reduction in Levels, at Least 1 Level, 2 Levels, and More Than 2 Levels of Improvement From Week 25 in Mobility, Self-care, and Usual Activities Domains of EQ-5D-5L
Description: EQ-5D-5L was assessed across 5 levels, with participants selecting the option that best described their health on that day, ranging from "no problems" to "unable to" walk, wash/dress, or perform usual activities. Out of total participants of each arm, only participants having no reduction, at least 1 Level, 2 Levels, and more than 2 Levels of improvement from baseline in Mobility, Self-care, and Usual Activities Domains of EQ-5D-5L are reported in this outcome measure.
Time Frame: From Week 25 to 41 and 53
Population: Analysis was performed on the mITT-Ex analysis set. The mITT-Ex comprised all participants in mITT who completed the first 24 weeks of SP1 and received any amount of the IMP in SP2. The documented failure to take any amount of randomized IMP in SP2 led to the exclusion of the participant from mITT-Ex. Here, overall number of participants analyzed (N) = participants evaluable for this outcome measure, and number analyzed (n) = participants with evaluable data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20
Number analyzed (Participants) | 47 | 45
Participants
  Week 41: Mobility: No Reduction | 29 | 28
  Week 41: Mobility: At least 1 level improvement | 10 | 8
  Week 41: Mobility: At least 2 level improvement | 1 | 0
  Week 41: Mobility: More than 2 level improvement | 0 | 1
  Week 41: Self-Care: No Reduction | 32 | 31
  Week 41: Self-Care: At least 1 level improvement | 5 | 9
  Week 41: Self-Care: At least 2 level improvement | 3 | 1
  Week 41: Self-Care: More than 2 level improvement | 0 | 0
  Week 41: Usual Activities: No Reduction | 23 | 31
  Week 41: Usual Activities: At least 1 level improvement | 13 | 10
  Week 41: Usual Activities: At least 2 level improvement | 1 | 1
  Week 41: Usual Activities: More than 2 level improvement | 1 | 0
  Week 53: Mobility: No Reduction: number analyzed (Participants) | 40 | 37
  Week 53: Mobility: No Reduction | 24 | 25
  Week 53: Mobility: At least 1 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Mobility: At least 1 level improvement | 8 | 7
  Week 53: Mobility: At least 2 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Mobility: At least 2 level improvement | 2 | 0
  Week 53: Mobility: More than 2 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Mobility: More than 2 level improvement | 0 | 1
  Week 53: Self-Care: No Reduction: number analyzed (Participants) | 40 | 37
  Week 53: Self-Care: No Reduction | 33 | 23
  Week 53: Self-Care: At least 1 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Self-Care: At least 1 level improvement | 2 | 11
  Week 53: Self-Care: At least 2 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Self-Care: At least 2 level improvement | 2 | 1
  Week 53: Self-Care: More than 2 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Self-Care: More than 2 level improvement | 0 | 0
  Week 53: Usual Activities: No Reduction: number analyzed (Participants) | 40 | 37
  Week 53: Usual Activities: No Reduction | 21 | 22
  Week 53: Usual Activities: At least 1 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Usual Activities: At least 1 level improvement | 10 | 10
  Week 53: Usual Activities: At least 2 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Usual Activities: At least 2 level improvement | 3 | 2
  Week 53: Usual Activities: More than 2 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Usual Activities: More than 2 level improvement | 0 | 0

31. Secondary Outcome: Percentage of Participants Having no Reduction in Levels, at Least 1 Level, 2 Levels, and More Than 2 Levels of Improvement From Week 25 in Mobility, Self-care, and Usual Activities Domains of EQ-5D-5L
Description: as for outcome 30
Time Frame: From Week 25 to 41 and 53
Population: as for outcome 30
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A: IgPro20 / IgPro20 | Sequence B: Placebo / IgPro20
Number analyzed (Participants) | 47 | 45
percentage of participants
  Week 41: Mobility: No Reduction | 61.7 | 62.2
  Week 41: Mobility: At least 1 level improvement | 21.3 | 17.8
  Week 41: Mobility: At least 2 level improvement | 2.1 | 2.2
  Week 41: Mobility: More than 2 level improvement | 0 | 0
  Week 41: Self-Care: No Reduction | 68.1 | 20.0
  Week 41: Self-Care: At least 1 level improvement | 0.6 | 20.0
  Week 41: Self-Care: At least 2 level improvement | 6.4 | 2.2
  Week 41: Self-Care: More than 2 level improvement | 0 | 0
  Week 41: Usual Activities: No Reduction | 48.9 | 68.9
  Week 41: Usual Activities: At least 1 level improvement | 27.7 | 22.2
  Week 41: Usual Activities: At least 2 level improvement | 2.1 | 2.2
  Week 41: Usual Activities: More than 2 level improvement | 2.1 | 0
  Week 53: Mobility: No Reduction: number analyzed (Participants) | 40 | 37
  Week 53: Mobility: No Reduction | 60.0 | 67.6
  Week 53: Mobility: At least 1 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Mobility: At least 1 level improvement | 20.0 | 18.9
  Week 53: Mobility: At least 2 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Mobility: At least 2 level improvement | 5.0 | 0
  Week 53: Mobility: More than 2 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Mobility: More than 2 level improvement | 0 | 2.7
  Week 53: Self-Care: No Reduction: number analyzed (Participants) | 40 | 37
  Week 53: Self-Care: No Reduction | 82.5 | 62.2
  Week 53: Self-Care: At least 1 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Self-Care: At least 1 level improvement | 5.0 | 29.7
  Week 53: Self-Care: At least 2 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Self-Care: At least 2 level improvement | 5.0 | 2.7
  Week 53: Self-Care: More than 2 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Self-Care: More than 2 level improvement | 0 | 0
  Week 53: Usual Activities: No Reduction: number analyzed (Participants) | 40 | 37
  Week 53: Usual Activities: No Reduction | 52.5 | 59.5
  Week 53: Usual Activities: At least 1 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Usual Activities: At least 1 level improvement | 25.0 | 27.0
  Week 53: Usual Activities: At least 2 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Usual Activities: At least 2 level improvement | 7.5 | 5.4
  Week 53: Usual Activities: More than 2 level improvement: number analyzed (Participants) | 40 | 37
  Week 53: Usual Activities: More than 2 level improvement | 0 | 0

32. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs), Related TEAEs and Serious TEAEs
Time Frame: Up to 5 years
Population: Period 1: Safety analysis set (SAF): All randomized participants who received any IMP, analyzed by actual treatment. Period 2: SAF extended (SAF-EX): Participants from SAF who completed 24 weeks in Period 1 and received any IMP in Period 2. Period 3: SAF for SP3 (SAF-P3): Participants from SAF-EX who completed 52 weeks in Periods 1 and 2 and received any IMP after Week 52.
Measure: Number; unit: percentage of participants
Groups:
- Period 1 Sequence A: IgPro20: Participants received IgPro20 SC infusions weekly for 24 weeks in Period 1.
- Period 1 Sequence B: Placebo: Participants received matching placebo SC infusions weekly for 24 weeks in Period 1.
- Period 2 Sequence A: IgPro20 / IgPro20: Participants received IgPro20 SC infusions weekly for 24 weeks in Period 1, followed by IgPro20 SC infusions weekly for 28 weeks in Period 2.
- Period 2 Sequence B: Placebo / IgPro20: Participants received matching placebo SC infusions weekly for 24 weeks in Period 1, followed by IgPro20 SC infusions weekly for 28 weeks in Period 2.
- Period 3 Sequence A: IgPro20/ IgPro20 / IgPro20: Participants received IgPro20 SC infusions weekly for 24 weeks in Period 1, followed by IgPro20 SC infusions weekly for 28 weeks in Period 2. At Week 53, participants with demonstrated treatment benefit at Week 49 (TIS >= 20 points) continued to Period 3 long-term treatment with open-label IgPro20 SC infusions weekly until the EOS (up to 5 years).
- Period 3 Sequence B: Placebo / IgPro20 / IgPro20: Participants received matching placebo SC infusions weekly for 24 weeks in Period 1, followed by IgPro20 SC infusions weekly for 28 weeks in Period 2. At Week 53, participants with demonstrated treatment benefit at Week 49 (TIS >= 20 points) continued to Period 3 long-term treatment with open-label IgPro20 SC infusions weekly until the EOS (up to 5 years).
Arm/Group | Period 1 Sequence A: IgPro20 | Period 1 Sequence B: Placebo | Period 2 Sequence A: IgPro20 / IgPro20 | Period 2 Sequence B: Placebo / IgPro20 | Period 3 Sequence A: IgPro20/ IgPro20 / IgPro20 | Period 3 Sequence B: Placebo / IgPro20 / IgPro20
Number analyzed (Participants) | 67 | 67 | 56 | 55 | 36 | 34
percentage of participants
  TEAEs | 82.1 | 67.2 | 69.6 | 74.5 | 75.0 | 76.5
  Related TEAEs | 52.2 | 25.4 | 17.9 | 43.6 | 13.9 | 20.6
  Serious TEAEs | 4.5 | 7.5 | 3.6 | 5.5 | 13.9 | 20.6

33. Secondary Outcome: Annualized Rate of TEAEs, Related TEAEs and Serious TEAEs Per Time at Risk
Time Frame: Up to 5 years
Population: Period 1: SAF: All randomized participants who received any IMP, analyzed by actual treatment. Period 2: SAF-EX: Participants from SAF who completed 24 weeks in Period 1 and received any IMP in Period 2. Period 3: SAF-P3: Participants from SAF-EX who completed 52 weeks in Periods 1 and 2 and received any IMP after Week 52.
Measure: Number; unit: TEAEs per year
Arm/Group | Period 1 Sequence A: IgPro20 | Period 1 Sequence B: Placebo | Period 2 Sequence A: IgPro20 / IgPro20 | Period 2 Sequence B: Placebo / IgPro20 | Period 3 Sequence A: IgPro20/ IgPro20 / IgPro20 | Period 3 Sequence B: Placebo / IgPro20 / IgPro20
Number analyzed (Participants) | 67 | 67 | 56 | 55 | 36 | 34
TEAEs per year
  TEAEs | 11.725 | 5.359 | 4.922 | 6.718 | 3.165 | 3.644
  Related TEAEs | 6.327 | 0.936 | 1.348 | 2.166 | 0.195 | 0.240
  Serious TEAEs | 0.214 | 0.226 | 0.067 | 0.110 | 0.137 | 0.288

34. Secondary Outcome: Annualized Rate of Mild, Moderate, and Severe TEAEs Per Time at Risk
Time Frame: Up to 5 years
Population: as for outcome 33
Measure: Number; unit: TEAEs per year
Arm/Group | Period 1 Sequence A: IgPro20 | Period 1 Sequence B: Placebo | Period 2 Sequence A: IgPro20 / IgPro20 | Period 2 Sequence B: Placebo / IgPro20 | Period 3 Sequence A: IgPro20/ IgPro20 / IgPro20 | Period 3 Sequence B: Placebo / IgPro20 / IgPro20
Number analyzed (Participants) | 67 | 67 | 56 | 55 | 36 | 34
TEAEs per year
  Mild | 9.151 | 4.035 | 4.011 | 4.332 | 2.442 | 2.157
  Moderate | 2.145 | 1.162 | 0.843 | 2.239 | 0.606 | 1.390
  Severe | 0.393 | 0.161 | 0.067 | 0.110 | 0.117 | 0.096

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Analysis was performed on the SAF, which consisted of all participants who were randomized and received any amount of randomized IMP and was based on the actual treatment sequence received.
Groups:
- Period 1 Sequence B: Placebo: Participants received albumin solution administered IV to match IgPro20 SC infusions weekly for 24 weeks in Period 1.
- Period 2 Sequence B: Placebo / IgPro20: Participants received albumin solution administered IV to match IgPro20 SC infusions weekly for 24 weeks in Period 1, followed by IgPro20 SC infusions weekly for 28 weeks in Period 2.
- Period 3 Sequence A: IgPro20/ IgPro20 / IgPro20: Participants received IgPro20 SC infusions weekly for 24 weeks in Period 1, followed by IgPro20 SC infusions weekly for 28 weeks in Period 2. At the Week 53 visit, eligible participants continued to study Period 3 and continued to receive IgPro20 SC infusions weekly until the end of the study.
- Period 3 Sequence B: Placebo / IgPro20 / IgPro20: Participants received albumin solution administered IV to match IgPro20 SC infusions weekly for 24 weeks in Period 1, followed by IgPro20 SC infusions weekly for 28 weeks in Period 2. At the Week 53 visit, eligible participants continued to study Period 3 and continued to receive IgPro20 SC infusions weekly until the end of the study.
Arm/Group | Period 1 Sequence A: IgPro20 | Period 1 Sequence B: Placebo | Period 2 Sequence A: IgPro20 / IgPro20 | Period 2 Sequence B: Placebo / IgPro20 | Period 3 Sequence A: IgPro20/ IgPro20 / IgPro20 | Period 3 Sequence B: Placebo / IgPro20 / IgPro20
All-Cause Mortality (participants affected / at risk) | 1/67 | 1/67 | 1/56 | 0/55 | 0/36 | 1/34
Serious Adverse Events (participants affected / at risk) | 3/67 | 5/67 | 2/56 | 3/55 | 5/36 | 7/34
Other Adverse Events (participants affected / at risk) | 41/67 | 33/67 | 25/56 | 33/55 | 21/36 | 17/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 Sequence A: IgPro20 (N=67) | Period 1 Sequence B: Placebo (N=67) | Period 2 Sequence A: IgPro20 / IgPro20 (N=56) | Period 2 Sequence B: Placebo / IgPro20 (N=55) | Period 3 Sequence A: IgPro20/ IgPro20 / IgPro20 (N=36) | Period 3 Sequence B: Placebo / IgPro20 / IgPro20 (N=34)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudolymphoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatomyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mueller's mixed tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 Sequence A: IgPro20 (N=67) | Period 1 Sequence B: Placebo (N=67) | Period 2 Sequence A: IgPro20 / IgPro20 (N=56) | Period 2 Sequence B: Placebo / IgPro20 (N=55) | Period 3 Sequence A: IgPro20/ IgPro20 / IgPro20 (N=36) | Period 3 Sequence B: Placebo / IgPro20 / IgPro20 (N=34)
Vertigo (Ear and labyrinth disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 5 (5) | 3 (3) | 2 (2) | 3 (6)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
Infusion site bruising (General disorders) | 5 (10) | 4 (10) | 1 (7) | 1 (1) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 12 (47) | 4 (4) | 1 (12) | 10 (11) | 0 (0) | 0 (0)
Infusion site nodule (General disorders) | 2 (2) | 0 (0) | 3 (6) | 1 (1) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 4 (10) | 1 (1) | 1 (1) | 5 (6) | 1 (2) | 0 (0)
Infusion site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (8) | 2 (2) | 0 (0)
Infusion site swelling (General disorders) | 6 (11) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (5)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 4 (4) | 6 (6) | 4 (4) | 13 (13) | 8 (8)
Cystitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 2 (9)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 5 (5) | 8 (21) | 6 (16)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 2 (3) | 2 (3) | 4 (8)
Fibrin D dimer increased (Investigations) | 5 (5) | 3 (4) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (2) | 4 (4) | 2 (3) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Dermatomyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (5) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (37) | 3 (3) | 3 (3) | 3 (4) | 4 (4) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 1 (1) | 2 (3) | 2 (3) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
A Good Clinical Practice (GCP) breach was identified and reported to regulatory authorities regarding insufficient safety information provided by one site for one Suspected Unexpected Serious Adverse Reaction (SUSAR) and one Adverse Event of Special Interest (AESI). The sponsor made repeated requests to obtain verification of the data, which the site did not provide. This limitation may have impacted the completeness of safety data characterization for these specific events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT04044690/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/90/NCT04044690/SAP_001.pdf